CLINICAL TRIAL: NCT07118657
Title: Host-Diet-Gut Interaction Post Vegan Diet in Pediatric Autoimmune Hepatitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AIH-03
Record Dates: First submitted 2025-05-08; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan Diet (Experimental)
  Interventions: Other: Vegan Diet
- Standard Diet (Active Comparator)
  Interventions: Other: Standard Diet

INTERVENTIONS:
Other: Vegan Diet — Vegan diet would be defined as a diet based solely of plant products with exclusion of all animal products including meat, fish, dairy, honey and eggs.• Additional supplementation of vitamin B12 (500 µg/day) in the vegan diet group along with calcium (50-75 mg/kg/day), vitamin D (800-1600 IU/day) and iron supplementation (3-6 mg/kg/day) as per requirement.
  o Monitoring- Based on vitamin B12 levels, 25(OH) vitamin D3 levels, serum calcium, and serum iron studies (complete hemogram, ferritin, iron, transferrin saturation, total iron binding capacity).
  Arms: Vegan Diet
Other: Standard Diet — Standard Diet
  Arms: Standard Diet

SUMMARY:
Pediatric autoimmune liver diseases (AILDs), including autoimmune hepatitis (AIH) and overlap syndromes like sclerosing cholangitis, are among the most common chronic liver conditions in the pediatric population. Currently, the treatment for AIH often involves long-term use of immunosuppressive therapy, which carries risks of severe side effects both in the short and long term. Due to these potential adverse effects, there is a critical need to explore alternative therapies that can modulate autoimmunity and potentially reduce or eliminate the dependence on immunosuppressive drugs. Autoimmune diseases, including AIH, typically arise in genetically predisposed individuals after exposure to certain environmental factors, leading to a breakdown in self-tolerance.The gut microbiome plays a crucial role in modulating the immune system through both anti-inflammatory and pro-inflammatory pathways. In advanced liver diseases, factors such as intestinal dysmotility, small intestinal bacterial overgrowth (SIBO), and increased intestinal permeability contribute to enhanced bacterial translocation, consistent with the "leaky gut" hypothesis. This phenomenon allows the passage of toxins, antigens, and bacteria into the systemic circulation, potentially exacerbating autoimmune responses. Consequently, altering the gut microbiome through dietary changes, probiotics, prebiotics, or fecal microbiota transplantation presents a promising therapeutic approach for autoimmune diseases.This study aims to investigate the gut microbiome and its modification following dietary intervention (specifically, a plant-based vegan diet) in pediatric AIH. Additionally, investigator will explore the potential role of such interventions in managing intestinal dysfunction in patients with advanced liver disease. In Aim 1, investigator will compare the baseline gut microbiome profiles of treatment-naïve pediatric AIH patients with those of healthy, age- and sex-matched controls to provide foundational insights. In Aim 2, investigator will evaluate the proportion of patients achieving biochemical remission after 180 days of a vegan versus standard diet in AIH patients. Investigator will also assess changes in stool metagenomics, metabolomics, cytokine profiles, gut epithelial barrier function, and liver disease severity scores between the two dietary groups.

This study aims to demonstrate the potential benefits of a vegan diet in managing autoimmune hepatitis. It seeks to provide evidence supporting dietary modifications as a complementary approach to standard medical treatments for a wide range of autoimmune or autoimmune-like disorders, potentially paving the way for future therapeutic strategies.

DETAILED DESCRIPTION:
Hypothesis/Research Question:

1. P = Population/Patient/Problem - Pediatric patients (< 18 years of age) with Autoimmune Hepatitis
2. I = Intervention -Vegan diet for 180 days (in addition of standard immunosuppressive medical therapy)
3. C = Comparison - Standard High Protein diet for 180 days (in addition of standard immunosuppressivemedical therapy)
4. O = Outcome - Proportion of subjects achieving biochemical remission; change in stool metagenome/metabolome/cytokines, gut epithelial barrier function, and liver disease severity scores between the two study groups.

Methodology:

Place: Department of Pediatric Hepatology &Molecular and Cellular Medicine, Institute of Liver and Biliary Sciences, New Delhi

* Study design: Prospective, Randomized, Single center, Open label study
* Study period: October 2024 to October 2027 Details of the diets (Vegan diet and Standard High Protein diet) Vegan diet would be defined as a diet based solely of plant products with exclusion of all animal products including meat, fish, dairy, honey and eggs.
* Additional supplementation of vitamin B12 (500 µg/day) in the vegan diet group along with calcium (50-75 mg/kg/day), vitamin D (800-1600 IU/day) and iron supplementation (3-6 mg/kg/day) as per requirement.

  * Monitoring- Based on vitamin B12 levels, 25(OH) vitamin D3 levels, serum calcium, and serum iron studies (complete hemogram, ferritin, iron, transferrin saturation, total iron binding capacity).

ELIGIBILITY:
Inclusion Criteria:

1. Cases diagnosed as Autoimmune hepatitis (AIH).
2. Controls are healthy subjects.

Exclusion Criteria:

1. Recent (< 6 weeks) exposure to oral or intravenous antibiotics, probiotics/prebiotics, proton pump inhibitors, or herbal medicines.
2. Any history of malignancy or any gastrointestinal tract surgery.
3. Recent (< 2 weeks) gastrointestinal infection.
4. Any dietary allergies .

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving biochemical remission after 180 days of vegan and standard high protein diet in treatment naive pediatric subjects with autoimmune hepatitis. | 180 days
  biochemical remission is defined as normalization of both serum AST/ALT & serum IgG.
  high protein (2-3 g/kg/day)

SECONDARY OUTCOMES:
Change in stool metagenome (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days
Change in stool metabolome (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days
Change in stool & blood cytokines (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days
Change in blood flow cytometry (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days
Change in Gut Epithelial Barrier Function (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days
Change in liver disease severity score (after 180 daysof plant based (vegan) vs. standard high protein diet along with standard medical management including immunosuppression in treatment naive pediatric subjects with autoimmune hepatitis). | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided